CLINICAL TRIAL: NCT02689375
Title: Rospective, Open Label, Pilot Study of Patient OutcoMes Following Successful TriAl of High Frequency SpInal CorD Stimulation at 10kHz (HF10™) Leading to Permanent Implant Compared to Trial Failure and Standard CarE for the TreatmeNt of Persistent Low BACK Pain of Neuropathic Origin
Brief Title: A Prospective, Open Label, Pilot Study of Patient OutcoMes Following Successful TriAl of High Frequency SpInal CorD Stimulation at 10kHz (HF10™) Leading to Permanent Implant Compared to Trial Failure and Standard CarE for the TreatmeNt of Persistent Low BACK Pain of Neuropathic Origin
Acronym: Maiden Back
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PM13/10904
Record Dates: First submitted 2015-02-11; First posted 2016-02-23 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients to receive spinal cord stimulator (Experimental)
  Interventions: Device: Senza Spinal Cord Stimulation system

INTERVENTIONS:
Device: Senza Spinal Cord Stimulation system — Suitable participants will be booked to have spinal cord stimulator trial leads implanted and an external programmable High Frequency battery trial box as a day case

SUMMARY:
25 participants with back pain and no previous spinal surgery will be enrolled from a single NHS site in England.

Participants will have already discussed spinal cord stimulation (SCS) pain management with their consultant before being invited to participate. Participants will attend for 10 visits over a period of 66 months. At visit one, study suitability screening and informed consent will be conducted. Suitable participants will be booked to have SCS trial leads implanted and an external programmable High Frequency battery trial box as a day case (Visit 2). Participants will be contacted over the next 21 days to assess how the trial is progressing and to book a follow up appointment in clinic to remove the trial leads (Visit 3) where a treatment decision will be made. If a participant is determined as having had a successful trial they will be listed and implanted with a full HF10 SCS implant (Visit 4). The participants who proceed to a full HF10 SCS implant will be reviewed in the Clinic at 6, 12, 24, 36, 48 and 60 months post procedure. Their participation in this study will be no longer than 66 months. A successful trial is defined as a reduction in pain by 30% on a Visual Analogue Scale. Participants who do not obtain 30% reduction in 21 days is classed as a failed trial and once the leads are removed will be reviewed in clinic by the investigator for an alternative treatment plan (Visit 4). If a participant is determined a failed trial of HF10, they will remain in the study with their consent for the full follow up schedule. The follow-up for the failed trial cohort can be conducted via telephone to reduce the burden on this trial group.

ELIGIBILITY:
Inclusion Criteria:

I. Patient is 18 years of age or older and has given written informed consent. II. Has persistent chronic predominant low back pain of neuropathic origin, with or with out radiculopathy, for a minimum of 6 months III. Visual Analogue Scale (VAS) back pain score of at least 50 mm at baseline IV. Confirmation of pain from neuropathic origin by SLANSS score (≥12) AND PainDETECT score( ≥19) V. Total daily dose of opioids equivalent to ≤200mg of Morphine VI. No previous open spinal surgery (percutaneous procedures such as nucleoplasty are not considered as open surgical procedures) VII. Failed conservative therapies such as physiotherapy, chiropractor, hydrotherapy, TENS.

VIII. MRI within the previous 18 months (as per standard care) IX. In the investigators opinion the patient is a suitable candidate for HF10

Exclusion Criteria:

I. Patient has mechanical spine instability based on flexion/extension testing of lumbar spine (documented in the last 6 months) II. Patient is pregnant, or pregnancy is suspected or planned within the first six months of the study timeframe.

III. Patient has a cardiac pacemaker, automatic defibrillator, or any other implanted device, which will make the trial impossible. IV. Allergy to device components or drugs to be used in the intended procedure. V. Medical co-morbidities that preclude surgical intervention. VI. Patient is incapable of understanding or responding to the study questionnaires VII. Patient is incapable of understanding or operating the patient programmer handset.

VIII. History of previous open spinal surgery (not percutaneous procedures) IX. Patient is morbidly obese (BMI ≥ 40). X. Patient is simultaneously participating in another device or drug study within the last 30 days.

XI. Patient has a spinal fracture, tumour or infection. XII. Clinical evidence of cauda equina syndrome. XIII. Progressive neurologic deficit.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-09-18 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
50% reduction in patient reported Visual analogue scale for pain | 12 months compared to baseline
50% reduction in patient reported numerical rating score for pain | 12 months compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom